CLINICAL TRIAL: NCT04482244
Title: Randomized, Double-blind Phase II Study of a Single Dose of Cannabidiol (CBD) for Acute Anticipatory Anxiety in Advanced Breast Cancer
Brief Title: RCT of CBD for Anxiety in Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Hans and Mavis Lopater Foundation (Unknown)
Responsible Party: Principal Investigator, Ilana Braun, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-886
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Advanced Breast Cancer; Anxiety; CBD
Keywords: Advanced Breast Cancer; Anxiety; CBD
MeSH Terms: conditions — Anxiety Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): After screening procedures confirm participation in the research study, participants will be randomized one of two groups:
  * Participants in the experimental arm will complete questionnaires and then receive a single dose of CBD prior to diagnostic CT scan or positron emission tomography (PET) .
  * Cannabidiol: Oral, per protocol dosage, single dose
  * Additional questionnaires 2 hours post scan and follow up via phone call 1 week regarding experience
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): After the screening procedures confirm participation in the research study, participants will be randomized one of two groups:
  * Participants in the placebo arm will complete questionnaire and then receive a single dose of placebo prior to diagnostic CT scan or positron emission tomography (PET) .
  * Placebo: Oral, per protocol dosage, single dose
  * Additional questionnaires 2 hours post scan and follow up via phone call 1 week regarding experience
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Liquid taken orally
  Other Names: Epidiolex; CBD
  Arms: Cannabidiol
Other: Placebo — Liquid taken orally
  Arms: Placebo

SUMMARY:
This research study is investigating use of a single dose of cannabidiol (CBD) to help manage anticipatory anxiety in participants with advanced breast cancer poised to undergo computed tomography (CT) or positron emission tomography (PET) to assess tumor burden.

The name of the study drug(s) are:

- Cannabidiol (CBD)

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Phase II trial of a single dose of CBD for acute anticipatory anxiety in patients with advanced breast cancer undergoing computed tomography (CT) or positron emission tomography (PET) to assess tumor burden.

The research study investigates use of CBD to manage anxiety prior to an oncologic imaging scan. CBD is a component of the cannabis sativa (marijuana) plant and of hemp. Studies of CBD have led to its approval by the Food and Drug Administration for certain childhood seizure disorders. Researchers have also been studying the use of CBD to manage anxiety and pain.

This study is designed to learn if the drug can help reduce anxiety and can safely be given to participants with advanced breast cancer who are scheduled for a CT or PET scan.

* After screening procedures confirm participation in the research study, participants will be "randomized" into one of two study groups: one group will receive CBD, the other group will receive a placebo of flavored corn syrup.
* Randomization means that participants are put into a group by chance. Neither the participant nor the research team will choose participant group assignment.

  * Participants will have a 66% chance of receiving a single dose of CBD.
  * Participants will have a 33% chance of receiving a single dose of placebo.
* On the day of treatment, participants will complete questionnaires before and after receiving a single dose of CBD or placebo then undergo computed tomography (CT) scan or positron emission tomography (PET). Participants will be contacted by phone approximately a week later and interviewed about study drug consumption and the CT/PET scan experience.

This study is supported by funding from the Hans and Mavis Lopater Foundation.

Approximately 50 people are anticipated to take part in this study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied. The FDA (the U.S. Food and Drug Administration) has not approved CBD to manage anxiety but it has been approved for use in children with some seizure disorders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stage IV or metastatic breast cancer
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%).
* Participants must have adequate organ and marrow function at baseline as defined below:

  * total bilirubin >2 times institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * Baseline anxiety as measured by GAD-7 ≥5
* At least mild anxiety typically experienced prior to oncologic scans (as measured by a prescreen survey item)

  * Computed tomography (CT) or positron emission tomography (PET) to assess tumor burden scheduled for within 48 hours of study drug administration
  * No cannabis, delta-9-tetrahydrocannabinol or cannabidiol use within 24-hours of study drug administration.
* No benzodiazepine consumption within 8 hours of study drug administration (e.g.,nighttime benzodiazepine use permissible)
* No driving for 12 hours following study drug administration.
* English proficiency
* The effects of cannabidiol (Epidiolex) on the developing human fetus are unknown. For this reason and because cannabis is known to be teratogenic, women of child-bearing potential must test as nonpregnant prior to entering the study. The study team will encourage women of child-bearing age and men to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 1 week after cannabidiol (Epidiolex) consumption. Women either age > 54 years or documented to be in menopause or status post hysterectomy will not be required to obtain bHCG.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cannabidiol (Epidiolex) or placebo (which contains sesame, corn and gluten)
* History of current clobazam or valproic acid use
* Current uncontrolled illness, for instance sepsis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
* Current use of antiretroviral therapy
* Participants with psychiatric illness or social situations that would limit compliance with study requirements
* Current hepatocellular carcinoma, or documented history of difficult to control diabetes -- Active participation in a clinical drug trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2026-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Braun, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Nayak MM, Chai P, Catalano PJ, Pirl WF, Tulsky JA, Tung SC, Lin NU, Andrade N, Johns S, Vaz C, Hughes M, Braun IM. Cannabidiol for Scan-Related Anxiety in Women With Advanced Breast Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2450391. doi: 10.1001/jamanetworkopen.2024.50391. PMID 39680411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the cancer center, medical records were screened between November 2, 2021, and March 1, 2023, and obtained physician approval prior to contacting potential participants. Interested women were consented and completed the survey and laboratory assessments necessary to determine eligibility. Survey assessments included demographics, cannabis history, the validated GAD-7 scale, and history of scan-related anxiety.
Pre-assignment Details: 501 screened. 310 excluded: 76 on clinical drug trial, 64 not responding, 37 declined,133 excluded for other reasons. Of 191 meeting eligibility, 54 without scheduled scan, 40 had scan too soon, 27 denied anxiety, & 3 excluded for other reasons. 67 scheduled for consent: 3 lost interest, 3 denied anxiety, & 1 did not attend. 60 patients consented, but 10 were not randomized, because they didn't meet eligibility criteria. 50 total participants were eligible, consented and randomized.
Groups:
- Cannabidiol: After screening procedures confirm participation in the research study, participants will be randomized one of two groups:
  * Participants in the experimental arm will complete questionnaires and then receive a single dose of CBD prior to diagnostic CT scan or positron emission tomography (PET) .
  * Cannabidiol: Oral, per protocol dosage, single dose
  * Additional questionnaires 2 hours post scan and follow up via phone call 1 week regarding experience
  Cannabidiol: Liquid taken orally
- Placebo: After the screening procedures confirm participation in the research study, participants will be randomized one of two groups:
  * Participants in the placebo arm will complete questionnaire and then receive a single dose of placebo prior to diagnostic CT scan or positron emission tomography (PET) .
  * Placebo: Oral, per protocol dosage, single dose
  * Additional questionnaires 2 hours post scan and follow up via phone call 1 week regarding experience
  Placebo: Liquid taken orally
Period: Overall Study
Arm/Group | Cannabidiol | Placebo
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cannabidiol | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Full Range); unit: years] | 60 [30 to 79] | 57 [37 to 81] | 58 [30 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 1
  Black of African American | 0 | 1 | 1
  Native Hawaiian or Pacific Islander | 0 | 1 | 1
  White | 24 | 19 | 43
  Multiracial | 1 | 2 | 3
  Declined | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
baseline anxiety score [Number; unit: participants]
  Mild to moderate | 22 | 22 | 44
  Severe | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety Score-Visual Analog Mood Scale (VAMs) Anxiety Subscale
Description: Afraid is a negative mood subscale on the VAMS. Each subscale involves a 0 (neutral face or lack of endorsement) to 100 mm (mood face of extreme endorsement) a horizontal line with each pole having an associated mood descriptor. A raw score is a measure of distance from the neutral face (0 mm) to where the participant marks their mood to be in the moment. A linear transformation of a raw score is converted to a T-score and calculated to have a mean of 50 and an SD of 10. The manual provides a T-score conversion table based on sex and age bracket (18-54 years and 55-94 years). A 20T-score (+/-) difference in either direction between a pre- and posttest scores is interpreted as a reliable change in mood, and those differing by more than 30T-score (+/-) is interpreted as both a reliable and a clinically significant relevant threshold for change in mood. A change score for a given mood was calculated based on using T-scores of post-drug administration minus the pre-drug.
Time Frame: 1 day of the drug administration pre-dose (T2) and 3 +/- 1 hour after drug administration (T3) up to 1 day
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 25 | 25
T-Score | -19.1 (15.4) | -15.0 (10.9)

2. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (PRO-CTCAE™) 5.
Description: Measured using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE™) and a qualitative assessment, patient-reported side effects and acceptability of taking oral CBD (versus placebo) for managing anticipatory anxiety.
Time Frame: 1 day of the drug administration pre-dose (T2) and 3 +/- 1 hour after drug administration (T3) up to 1 weeks post ingestion
Measure: Count of Participants; unit: Participants
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 25 | 25
Participants | 2 | 0

3. Secondary Outcome: Change in Mood Score-Visual Analog Mood Scale (VAMs) Anxiety Subscale
Description: Confused, Sad, Angry, Tired, Tense are negative moods and Energetic and Happy are positive moods on VAMS. Each subscale involves a 0 (neutral face) to 100 mm (mood face) a horizontal line with each pole having an associated mood descriptor. A raw score is a measure of distance from the neutral face (0 mm) to where the participant marks their mood to be in the moment. A linear transformation of a raw score is converted to a T-score and calculated to have a mean of 50 and SD of 10. The manual provides a T-score conversion table based on sex and age bracket (18-54 years and 55-94 years). A 20T-score (+/-) difference in either direction between a pre- and posttest scores is interpreted as a reliable change in mood, and those differing by more than 30T-score (+/-) is interpreted as both a reliable and a clinically significant relevant threshold for change in mood. A change score for a given mood was calculated based on using T-scores of post-drug administration minus the pre-drug.
Time Frame: Baseline through 3 +/- 1 hour after drug administration (T3) up to 1 day
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 25 | 25
T-Score
  Confused | 0.9 (6.7) | -0.1 (4.9)
  Sad | -5.8 (11.2) | -8.9 (11.4)
  Angry | -3.6 (8.8) | -6.1 (10.5)
  Energetic | -1.8 (8.7) | -2.1 (13.6)
  Tired | -2.0 (9.8) | -3.6 (10.1)
  Happy | 3.3 (8.7) | 2.6 (9.3)
  Tense | -11.6 (12.6) | -10.4 (8.8)

4. Secondary Outcome: Nausea Rate
Description: Nausea and vomiting were measured using two items. Scale scores were calculated by averaging items within scales and transforming average scores linearly. All of the scales range in score from 0 to 100. A high score for a symptom scale or item represents a high level of symptomatology or problems.
Time Frame: Baseline through 3 +/- 1 hour after drug administration (T3) up to 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale
  NV Score Pre-drug | 6.0 (8.2) | 6.7 (13.6)
  NV Score Post-drug | 7.3 (15.3) | 1.3 (4.6)

5. Secondary Outcome: Numeric Pain Rating Scale (NPRS)
Description: pain intensity scale is scored from 0 to 10 (with 10 representing "worst possible" pain).
Time Frame: Baseline , 1 day of the drug administration pre-dose
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cannabidiol | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | -0.88 (1.45) | -0.88 (1.33)

ADVERSE EVENTS:
Time Frame: 1 week follow up
Arm/Group | Cannabidiol | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 2/25 | 0/25
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cannabidiol (N=25) | Placebo (N=25)
Pain (General disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
it excluded men, so its findings cannot be extrapolated beyond women.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/44/NCT04482244/Prot_SAP_000.pdf